CLINICAL TRIAL: NCT03428711
Title: Mesoglycan (Prisma®) Versus Placebo in Secondary Prevention of the Superficial Venous Thrombosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Quovadis Associazione (Other)
Collaborators: Neopharmed Gentili S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: METRO
Record Dates: First submitted 2018-01-30; First posted 2018-02-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Superficial Venous Thrombosis of Leg, Secondary Prevention
Keywords: Superficial Venous Thrombosis of Leg; secondary prevention; prophylaxis
MeSH Terms: interventions — mesoglycan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Oral Tablet (Placebo Comparator): Placebo comparator twice-a-day, for 12 months
  Interventions: Drug: Placebo Oral Tablet
- Mesoglycan Oral Tablet (Experimental): a mixture of glycosaminoglycans (mainly heparan-sulphate, dermatan sulfate), inhibitors of thrombin and of Factor Xa and active in restore flow-mediated vasodilation.
  50 mg, twice-a-day, for 12 months
  Interventions: Drug: Mesoglycan Oral Tablet

INTERVENTIONS:
Drug: Mesoglycan Oral Tablet — Experimental drug: mesoglycan, already used in the treatment of chronic venous ulcers, is a complex mucopolysaccharide, composed of a mixture of glycosaminoglycans (mainly heparan-sulphate, dermatan sulfate), inhibitors of thrombin and of Factor Xa and active in restore flow-mediated vasodilation.
  Used in oral formulation, hard capsules, 50 mg, twice-a-day, for 12 months. Reference therapy: placebo, organoleptically indistinguishable from the experimental drug, twice-a-day, for 12 months.
  Other Names: Prisma
  Arms: Mesoglycan Oral Tablet
Drug: Placebo Oral Tablet — Indistinguible placebo tablet
  Other Names: placebo
  Arms: Placebo Oral Tablet

SUMMARY:
The objective of the study is to demonstrate the superiority of the mesoglycan (Prisma®), compared to placebo, in reducing the incidence of thromboembolic complications (relapse / extension of superficial venous thrombosis (SVT), deep venous thrombosis (DVT), pulmonary embolism (PE)) in patients who have completed the cycle of therapy of the acute phase after superficial vein thrombosis.

DETAILED DESCRIPTION:
Rationale: SVT is a relatively common clinical condition, with recent evidence of association with the development of DVT and / or pulmonary embolism that has changed the perception of the risk of this disease (with conflicting data in the literature: 3-33 %). Previous natural history studies have observed that thromboembolic complications (relapse / extension of SVT, DVT, PE) can affect up to 10-15% of subjects at 3-6 months from the initial event, despite adequate treatment of the acute phase. There are no literature studies that have prospectively investigated the usefulness of drug therapy in secondary prevention of SVT once the initial therapeutic cycle is completed.

Objective: To demonstrate the superiority of the mesoglycan (Prisma®), compared to placebo, in reducing the incidence of thromboembolic complications (relapse / extension of superficial venous thrombosis (SVT), deep venous thrombosis (DVT), pulmonary embolism (PE)) in patients who have completed the cycle of therapy of the acute phase after superficial vein thrombosis.

Investigators: 18 Italian centers with proven experience in the treatment and prevention of venous thromboembolic disease.

Study Design:

Phase II, multicentre, randomized, double-blind superiority study comparing mesoglycan (Prisma®) 50 mg and placebo, both in double oral daily intake.

Study treatment:

Experimental drug: mesoglycan (Prisma®), already used in the treatment of chronic venous ulcers, is a complex mucopolysaccharide, composed of a mixture of glycosaminoglycans (mainly heparan-sulphate, dermatan sulfate), inhibitors of thrombin and of Factor Xa and active in restore flow-mediated vasodilation.

Used in oral formulation, hard capsules, 50 mg, twice-a-day, for 12 months. Reference therapy: placebo, organoleptically indistinguishable from the experimental drug, twice-a-day, for 12 months.

Masking: the study is conducted in "double-blind".

Methodology and phases of the study:

Written Consent Collection: the investigator will inform the interested party that participation in the study is voluntary and that the refusal will not lead to the loss of any benefit or in any way affect the relationship with the doctor. Furthermore, it will be announced that withdrawal from the study is possible at any time without having to provide a specific reason. Before being enrolled in the study, each subject will receive a complete explanation of the nature and purpose of the study by the investigator, along with a description of the benefits and risks associated with participation. Insurance coverage will also be mentioned and related procedures in case of injuries will be explained. A clear information sheet will be delivered to the subject covering all the important aspects of the study. Once read, the subject will have the opportunity to ask questions and sufficient time will be given to consider the various aspects presented, before being asked to sign and date the informed consent form.

The original copy of the signed and dated informed consent form will be kept by the investigator in the "study file" kept in the Center. The subject will receive a copy of the informed consent form signed and dated for future reference.

Screening: after obtaining written informed consent, all potential subjects will complete the screening visit. If they satisfy the prefixed inclusion and exclusion criteria, they will be enrolled in the study and will be subjected to ultrasound study using by color-coded duplex ultrasonography (CCDU) of the lower limbs (investigation in standard clinical practice because at the end of the treatment of the acute phase), to exclude a concomitant involvement of the deep venous circle, or an extension of the initial SVT, which would imply the extension of parenteral anticoagulant therapy. A blood test will be performed to determine complete blood count, ALT, AST, creatinine, PT-INR, aPTT and PCR.

Randomization: centralized, through a specific application of the EDC website, with 1: 1 allocation (stratified by age <60 /> = 60 years old and gender, in blocks of variable size, random of 4 and 6 units) between placebo and mesoglycan. It is estimated that enrollment was completed in 24 months.

Scheduled visits: check-ups at 3, 6, 9, 12 months during treatment and at 24 months with:

* overall clinical evaluation and treatment compliance,
* collection of information on any thromboembolic events and / or adverse events,
* evaluation of rVCSS and VEINES / Sym-QoL scores,
* at 12 months, CCDU and blood sampling for complete blood counts, ALT, AST, creatinine, PT-INR, aPTT and PCR.
* at 24 months, blood sampling for complete blood counts, ALT, AST, creatinine, PT-INR, aPTT and PCR.

The subject will be instructed to be present at any time for a clinical check in case of signs / symptoms suggestive of thromboembolic events.

During the treatment period on days: 30, 60, 135, 225, 315 (+ -5 days) from the randomization, and in the follow-up period after 3, 6 and 9 months from the end of the treatment and then every 6 months until the end of the study, the subjects will be contacted by telephone by trained personnel to assess their compliance with treatment, the possible use of drugs not allowed and the onset of adverse events and / or end-points of the study.

The concomitant use of oral or parenteral anticoagulants, phlebotropics, NSAIDs in chronic and continuous treatment (except for the occasional symptomatic use of NSAIDs), double-anti-aggregation or ASA> 160 mg / day, centrally acting painkillers is not permitted during the study.

The contemporary use of elasto-compressive therapy, of which there is no evidence of real effectiveness, is left to the clinician's judgment.

Participants will exit permanently from the study if it occurs: one of the primary end-points, the onset of one of the exclusion criteria, a serious adverse event (SAE) that achieves one of the exclusion criteria, the withdrawal of consent.

Evaluation criteria:

Primary efficacy end-point: Cumulative occurrence of the first event, with instrumental confirmation, occurring during the study treatment between: recurrence or extension of, asymptomatic or symptomatic, SVT, new DVT (proximal asymptomatic or symptomatic / symptomatic isolated distal), pulmonary embolism (fatal or symptomatic non-fatal).

Secondary efficacy end-points: Cumulative occurrence of the first event between: recurrence or extension of, asymptomatic or symptomatic, SVT, new proximal / distal DVT (asymptomatic or symptomatic), pulmonary embolism (fatal or symptomatic non-fatal); modification of the rVCSS score (efficacy) and VEINES / Sym-QoL (quality of life) in treatment and in the following 12 months; recanalization of the vein involved in the primary thrombotic event; new development of deep and / or superficial venous reflux; impact of elasto-compressive therapy; contribution of PCR levels in predicting the onset of the primary end-point.

Security End-Point: Serious adverse events, Total adverse events. Hemorrhagic AEs are classified as major or minor (ISTH Guidelines).

A copy of the Diagnostic Report of the first event considered will be compulsorily collected and transmitted to the coordinating center for the validation of the event.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of both genders, aged> = 18 years,
2. With previous diagnosis of SVT of the lower limbs documented by color-coded duplex ultrasonography (CCDU), which at the onset was at least 5 cm of extension and at least 3 cm from the saphenous junctions (vena magna saphenous and saphenous),
3. who have completed the initial therapeutic cycle with Fondaparinux 2.5 mg / day for 45 days, as required by the most recent Guidelines (ACCP).
4. That screening CCDU does not show deep venous involvement, or an extension of the initial SVT.

Exclusion Criteria:

1. Poor compliance with the treatment of SVT,
2. life expectancy <24 months,
3. anticipated lack of cooperation or impossibility to complete the questionnaires,
4. pregnancy, lactation or programmed pregnancy during the duration of the study,
5. severe locomotor disability or prolonged immobilization,
6. participation in another study in the last 3 months,
7. post-thrombotic syndrome with "Villalta score"> 4,
8. chronic lymphedema of the lower limbs,
9. recent (<3 months) or planned interventional drip-surgery or trans-luminary arterial percutaneous angioplasty (PTA),
10. ongoing dialysis treatment,
11. malabsorption / malnutrition status,
12. chronic and non-suspendable use of anticoagulants, phlebotropics, corticosteroids or NSAIDs, double-antiaggregation or ASA> 160mg / die, centrally acting painkillers,
13. subjects with hypersensitivity to the mesoglycan, heparin or heparinoids, intolerant to galactose or with lactase deficiency, carriers of hemorrhagic diathesis or diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Cumulative thrombosis recurrence | 12 months
  Cumulative occurrence of the first event, with instrumental confirmation, occurring during the study treatment between: recurrence or extension of, asymptomatic or symptomatic, SVT, new DVT (proximal asymptomatic or symptomatic / symptomatic isolated distal), pulmonary embolism (fatal or symptomatic non-fatal).

SECONDARY OUTCOMES:
Cumulative thrombosis recurrence with distal | 12 months
  Cumulative occurrence of the first event between: recurrence or extension of, asymptomatic or symptomatic, SVT, new proximal / distal DVT (asymptomatic or symptomatic), pulmonary embolism (fatal or symptomatic non-fatal)
Symptoms | 12 months
  variation during the follow-up of the "revised Venous Clinical Severity Score" (rVCSS); min-max scale value 0-30; higher value represent a worse severity outcome.
VEINES-QOL/ Sym score | 12 months
  variation during the follow-up of the "Venous Insufficiency Epidemiological and Economic Study" (VEINES)-QOL/ Sym scores;
  subscale QOL: a venous disease-specific measure of quality of life; min-max scale value 0-100; higher value represent a better quality of life outcome.
  subscale Sym: a venous disease-specific measure of symptoms ; min-max scale value 0-100; higher value represent a better symptomatic outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Camporese, MD, Principal Investigator — Quovadis Associazione
Locations (1):
- Giuseppe Camporese, Padua, Padova, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camporese G, Bernardi E, Bortoluzzi C, Noventa F, Simioni P; METRO Investigator Study Group. Mesoglycan for the secondary prevention of superficial vein thrombosis: a randomized, controlled, double-blind study (METRO Study)-rationale and protocol. J Thromb Thrombolysis. 2024 Feb;57(2):226-234. doi: 10.1007/s11239-023-02896-6. Epub 2023 Nov 6. PMID 37932589